CLINICAL TRIAL: NCT02815111
Title: Evaluation of Ketamine and Multi-modal Analgesics for Postoperative Analgesia, Opioid Sparing, and Early Extubation in ICU Compared With Conventional Analgesia
Brief Title: Evaluation of Ketamine and Multi-modal Analgesics
Status: Withdrawn | Type: Observational
Why Stopped: Not IRB approved
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201600316
Record Dates: First submitted 2016-06-16; First posted 2016-06-28 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Ketamine; Lidocaine; Acetaminophen; Gabapentin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control Group: Intensivists will proceed with analgesia utilizing conventional opioid based pain order sets.
- Study Group: The investigators plan to study an analgesic regimen of Ketamine and lidocaine as infusions with Neurontin and Acetaminophen delivered orally for postoperative analgesia and the subsequent effect on ventilator days and ICU stay.
  Interventions: Drug: Ketamine; Drug: Lidocaine; Drug: Acetaminophen; Drug: Neurontin

INTERVENTIONS:
Drug: Ketamine — Receive an analgesic regimen that involves Ketamine infusions
  Other Names: Ketalar
  Groups: Study Group
Drug: Lidocaine — Receive an analgesic regimen that involves Lidocaine infusions
  Other Names: Lidopen
  Groups: Study Group
Drug: Acetaminophen — May be administered Acetaminophen rectally, by mouth, or intravenously in patients not suitable for either of the other methods of administration
  Other Names: Tylenol
  Groups: Study Group
Drug: Neurontin — May be given Neurontin by mouth as an approved medication for pain control
  Other Names: Gabapentin
  Groups: Study Group

SUMMARY:
The purpose of this research study is to see if pain can be better controlled with fewer side effects. The new drug regimen will study several different medicines that have different ways of treating pain.

DETAILED DESCRIPTION:
The investigators plan to study an analgesic regimen of Ketamine and Lidocaine as infusions with Neurontin and acetaminophen delivered orally for postoperative analgesia and the subsequent effect on ventilator days and ICU stay. The investigators expect that pain scores will be either unchanged or better than historic controls. In addition, the investigators expect that ventilator days and ICU stay will be improved due to reduced incidence of delirium and bowel dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) status 1-4
* Undergoing planned surgery for cardiac problems
* 18 years of age and not older than 85 years of age

Exclusion Criteria:

* Severe liver disease (alanine aminotransferase (ALT) , aspartate aminotransferase (AST), or bilirubin > 2.5 times Upper Limit of Normal)
* Pregnancy or currently breastfeeding
* History of schizophrenia or other hallucinatory psychiatric disorder
* History of chronic or pre-existing pain disorder
* History of heart block
* Severe renal impairment Creatinine Clearance (CrCl)<30 milliliter(mL)/min

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing planned surgery for cardiac problems
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2018-01 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Changes between the two groups assessed by overall ventilator days | Through study completion, an average of one week
  Total ventilator days

SECONDARY OUTCOMES:
Changes between the two groups assessed by ICU length of stay | Through study completion, an average of one week
  ICU length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Sean Kiley, M.D., Principal Investigator — University of Florida

IPD SHARING:
Plan to Share IPD: No